CLINICAL TRIAL: NCT02784470
Title: Study of Gastroduodenal Metallic Stent vs Gastrojejunostomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Moon-Won Yoo, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20151141
Record Dates: First submitted 2016-05-19; First posted 2016-05-27 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- gastrojejunostomy arm (Experimental)
  Interventions: Procedure: gastrojejunostomy
- gastroduodenal stent placement (Active Comparator)
  Interventions: Device: gastroduodenal stent placement

INTERVENTIONS:
Device: gastroduodenal stent placement
  Arms: gastroduodenal stent placement
Procedure: gastrojejunostomy
  Arms: gastrojejunostomy arm

SUMMARY:
Selection of the optimal treatment for gastric outlet obstruction in patients with radically unresectable gastric cancer remains controversial because previous studies comparing the two procedures had a small sample size as well as they included various etiologies such as gastrointestinal (GI) cancer, duodenal cancer and pancreaticobiliary cancer in selecting the patient population. Therefore, to establish the standard of care for patients with radically unresectable gastric cancer with gastric outlet obstruction, a larger prospective, randomized, controlled clinical trial using a single type of stent is warranted.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥19 to 80 years
* ECOG performance status 0-3
* Life expectancy >3 months
* Patients with malignant gastric outlet obstruction (distal part of stomach, pyloric ring or duodenal bulb obstruction) caused by gastric cancer
* Patients who are not eligible for radical operation due to local progression of gastric cancer, distant metastasis or his/her general condition.
* Patients with GOOSS score 0-2
* Patients with symptoms consistent with gastric outlet obstruction including persistent nausea and vomiting
* Patients with findings consistent with malignant gastric outlet obstruction on imaging studies including upper GI endoscopy, upper GIseries or abdominal computed tomography (CT)
* Patients who are eligible to undergo both gastroduodenal stent placement and gastrojejunostomy (eligibility will be determined by agreement by at least one gastroenterological surgeon and at least one radiologist)
* Patients who have been provided with an explanation of the procedures of the clinical trial, voluntarily decided participation and signed the informed consent form

Exclusion Criteria:

* Pregnant or lactating women
* Women of childbearing potential with positive pregnancy test at baseline. Post-menopausal women should have at least 12 months of amenorrhea to be considered not of childbearing potential.
* Patients who have previously undergone balloon dilatation or stent placement for malignant gastric outlet obstruction
* Patients with past history of palliative bypass surgery or gastrectomy
* Patients with peritoneal metastasis or multiple intestinal obstruction caused by other cause on imaging scan including abdominal CT or small bowel series
* Patients who have been treated for intestinal adhesion caused by previous abdominal surgery
* Patients who are not eligible for general anesthesia due to poor general condition
* Patients with clinical evidence of intestinal perforation or peritonitis
* Patients who are determined to be not eligible for stent placement or gastrojejunostomy due to other cause

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Gastric Outlet Obstruction Scoring System (GOOSS) score | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yoomoon Won, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea